CLINICAL TRIAL: NCT05888207
Title: A Phase I, Open-label, Fixed-sequence Study to Assess the Effects of Strong CYP1A2 Inhibitor (Fluvoxamine) on Savolitinib Exposure in Healthy Male Subjects
Brief Title: A Study to Assess the Effects of Fluvoxamine on Savolitinib Exposure in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: D5084C00015
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Healthy Male Subjects
Keywords: Fixed-sequence; CYP1A2 inhibitor; Drug-drug interaction
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Savolitinib/Savolitinib+Fluvoxamine (Experimental): In period 1, subjects will receive a single oral dose of savolitinib on Day 1 after overnight fasting. Following minimum 10 days of washout after the last dose of savolitinib, in period 2 subjects will take oral doses of fluvoxamine alone, twice daily from Days 1 to 4. On Day 5 subject will receive a single oral dose of savolitinib and a twice daily oral dose of fluvoxamine. On Day 6, subjects will receive a twice daily oral dose of fluvoxamine alone.
  Interventions: Drug: Savolitinib; Drug: Fluvoxamine

INTERVENTIONS:
Drug: Savolitinib — Savolitinib will be administered as a single oral dose on Day 1 of Period 1 and on Day 5 of Period 2.
Drug: Fluvoxamine — Only fluvoxamine will be administered as a twice daily oral dose from Days 1 to 4 of Period 2. On Day 5 of Period 2, subject will receive a twice daily oral dose of fluvoxamine along with savolitinib. On Day 6 of Period 2, subject will receive a twice daily oral dose of fluvoxamine alone.

SUMMARY:
This study will assess the effects of strong CYP1A2 (Cytochrome P450 1A2) inhibitor (fluvoxamine) on savolitinib exposure in healthy male subjects, performed at a single clinical unit.

DETAILED DESCRIPTION:
This study will be a Phase I, open-label, fixed-sequence, 2-treatment period study.

The study will consist of 2 periods. During period 1 of the study, each subject will receive a single oral dose of savolitinib following an overnight fast. A low-fat breakfast will be provided prior to dosing. There will be a minimum washout period of 10 days (14 days between two successive savolitinib doses) between period 1 and period 2.

During period 2 of the study, subject will take oral doses of fluvoxamine alone from Days 1 to 4. There would be no dietary restrictions for fluvoxamine dosing. On Day 5, subjects will take a single oral dose of savolitinib and oral dose of fluvoxamine. On Day 6, subject will receive an oral dose of fluvoxamine alone. Each subject would be involved in the study for 9 weeks (including screening window).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with suitable veins for cannulation or repeated venipuncture.
* Male subjects must use barrier contraception.
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Regular bowel movements.

Exclusion Criteria:

* History of any clinically significant disease or disorder, which in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, vital signs, 12 lead ECG and physical examination.
* QTcF > 450 ms or QT > 500 ms or other ECG abnormality making interpretation more difficult, as judged by the investigator, or a history of additional risk factors for Torsades de Points, which in the opinion of the investigator may put the subject at risk.
* Any positive result on screening for serum hepatitis B surface antigen OR anti-HBc antibody, indicative of active hepatitis B, hepatitis C antibody, or HIV antibody.
* History of latent or chronic infections.
* Known or suspected drug or alcohol abuse or positive drugs of abuse test. History of excessive alcohol assumption or chronic alcohol induced disease. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 1 month (30 days) of Visit 2 (Day -1 of Period 1) or 5 half lives whichever longer in this study or participation in a method development study (no drug) 1 month prior to Visit 2. The period of exclusion begins 1 month after the final dose or 5 half-lives after the final dose or 1 month after the last visit, whichever is the longest.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 6 months prior to screening.
* Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies (which include but are not limited to: kava, ephedra [ma hung], ginko biloba, dehydroepiandrosterone, yohimbe, saw palmetto and ginseng), megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer (> 5 half-lives) if the medication has a long half-life.
* Subject has clinical signs and symptoms consistent with COVID-19, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission unless confirmed by a negative SARS CoV-2 PCR test.
* History of severe COVID-19 (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).
* Excessive intake of caffeine-containing drinks or food.
* Planned in-patient surgery, dental procedure, or hospitalization during the study.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug.
* Received a seasonal flu vaccine (including H1N1, H1N5) 28 days prior to first dose of study drug.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) for savolitinib | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the effects of fluvoxamine on savolitinib Cmax in healthy male subjects after administration of a single oral dose.
Area under plasma concentration time curve from zero to infinity (AUCinf) for savolitinib | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the effects of fluvoxamine on savolitinib AUCinf in healthy male subjects after administration of a single oral dose.

SECONDARY OUTCOMES:
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) for savolitinib | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the AUClast of savolitinib when administered alone or in combination with fluvoxamine.
AUClast for metabolites M2 and M3 | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the AUClast of savolitinib metabolites (M2 and M3) when savolitinib is administered alone or in combination with fluvoxamine.
Cmax for metabolites M2 and M3 | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the Cmax of savolitinib metabolites (M2 and M3) when savolitinib is administered alone or in combination with fluvoxamine.
AUCinf for metabolites M2 and M3 | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the AUCinf of savolitinib metabolites (M2 and M3) when savolitinib is administered alone or in combination with fluvoxamine.
Ratio of metabolite Cmax to parent Cmax (MRCmax) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the MRCmax of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Ratio of metabolite AUCinf to parent AUCinf (MRAUCinf) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the MRAUCinf of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Ratio of metabolite AUClast to parent AUClast (MRAUClast) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the MRAUClast of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) for savolitinib and metabolites (M2 and M3) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the tmax of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t1/2λz) for savolitinib and metabolites (M2 and M3) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the t1/2λz of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Terminal rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz) for savolitinib and metabolites (M2 and M3) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the λz of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Number of data points used for λz determination (λzN) for savolitinib and metabolites (M2 and M3) | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the λzN of savolitinib and its metabolites (M2 and M3) when savolitinib is administered alone.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) for savolitinib | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the CL/F of savolitinib when savolitinib is administered alone.
Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) for savolitinib | Period 1: Day 1 to Day 3 and Period 2: Day 5 to Day 7
  To evaluate the Vz/F of savolitinib when savolitinib is administered alone.
Number of subjects with adverse events (AEs) | From screening (Day -28 to Day -2) to follow up visit (approximately 9 weeks)
  To assess additional safety and tolerability of savolitnib.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home